CLINICAL TRIAL: NCT01221389
Title: Study Using Plasma for Patients Requiring Emergency Surgery: A Randomized Pilot Trial of Early Plasma for Patients Undergoing Emergency Surgery for Hemorrhagic Shock
Brief Title: Study Using Plasma for Patients Requiring Emergency Surgery
Acronym: SUPPRES
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding to afford plasma
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Dave Neilipovitz, Physician, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: OHREB#2010077-01H
Record Dates: First submitted 2010-08-19; First posted 2010-10-15 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Hemorrhagic Shock; Blood Coagulation Disorders; Blood Products; Trauma; Ruptured AAA
Keywords: hemorrhage; plasma; coagulopathy; trauma
MeSH Terms: conditions — Shock, Hemorrhagic; Blood Coagulation Disorders; Wounds and Injuries; Hemorrhage; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colloid Control (Active Comparator): Patients will receive 2 units of 250 ml of hydroxyethylated starch solution once they are sent to the OR for emergency surgery to address etiology for hemorrhagic shock.
  Interventions: Drug: Human Plasma
- Plasma (Active Comparator): Patients will receive 2 units of AB+ plasma once they are sent to the OR for emergency surgery to address etiology for hemorrhagic shock.
  Interventions: Drug: Human Plasma

INTERVENTIONS:
Drug: Human Plasma — Patients will receive either 2 units of AB+ plasma or 2 units of hydroxyethylated starch control solution once they are sent to the OR for emergency surgery to address etiology for hemorrhagic shock.
  Other Names: non applicable

SUMMARY:
Information on the management of casualties from the ongoing conflicts in Afghanistan and Iraq has brought in to question the traditional approach to blood transfusion in hemorrhaging patients. Present recommendations for when to transfuse plasma products is when coagulation tests become abnormal. The proposed trial will investigate whether the more aggressive plasma transfusion strategies as advocated from researchers based on the Central Asian conflicts is valid. Since a study to determine the full impact of an altered plasma transfusion practice would require thousands of patients, a feasibility trial is appropriate and is being proposed. The hypotheses are thus:

Primary Hypothesis- A multicentre trial that investigates the earlier use of plasma in patients with hemorrhagic shock going for emergency surgery will be feasible.

Secondary Hypotheses- The early use of a universal donor blood plasma (AB+ plasma) in patients with shock due to blood loss (i.e. hemorrhagic) going for emergency surgery will reduce overall exposure to the total number of blood donor products (so-called allogeneic blood exposure). A reduction in allogeneic blood exposure would then reduce the total number of blood transfusion-related complications. The early use of this plasma product is safe and will not increase the incidence of blood clotting or other transfusion-related complications.

DETAILED DESCRIPTION:
Investigations that have arisen from reviews of casualty management in the ongoing conflicts in Afghanistan and Iraq have challenged the standard approach to blood transfusion in hemorrhaging patients. Present recommendations are to ideally transfuse non-red blood cell blood products as indicated by coagulation and other blood tests. In the event that testing is not available or feasible, then clinical judgment is advised with two recommendations. The first is that platelets are usually required after red blood cell (RBC) transfusions of one blood volume (approximately 5 liters of blood loss); and the second is that plasma is not usually required until RBC transfusion of well over one blood volume. Contrary to these recommendations is evidence from these conflicts indicating that delays in plasma transfusion or reduced plasma dosing are associated with increased mortality. Although the evidence is primarily retrospective and at times circumstantial in nature, the relationship between plasma administration and mortality appears to be causation rather than simple association. Matching of injury severity and other important variables does not alter this conclusion. If this conclusion is true, the question becomes whether or not the transfusion practice of patients in a civilian setting should be changed.

The present plasma transfusion recommendations were largely based on studies of plasma exchange patients and the use of data from the 1970's. In plasma exchange, patients have a controlled removal of their plasma that is ultimately replaced with donor plasma. Coagulopathy develops solely from the amount of plasma removal since no consumption of factors exists. Hemorrhaging patients however lose coagulation factors both in shed blood and due to ongoing consumption at sites of injury. Further, the hemodynamic instability and hypovolemia experienced by hemorrhaging patients further exacerbates the reduction in clotting factor levels. Prior to the late 1980's, hemorrhaging patients often received whole blood transfusions. Whole blood, no longer used in most circumstances, contains approximately 1 unit of plasma in each unit. Thus, patients receiving whole blood will not develop a coagulopathy as quickly as patients who receive the now standard packed red blood cell units.

Despite a lack of prospective studies and significant limitations of the supporting evidence, the practice of waiting to administer plasma was rapidly adopted. Reasons for this were several but included concerns about infectious transmissions, shortage of blood products and the financial costs of the blood products. Regardless of the reasons for their development however, the present transfusion recommendations including those for plasma may no longer be applicable in all circumstances.

A strong argument against waiting for the coagulopathy to develop before treating is that the consequences of the coagulopathy are so grave that they should be avoided. The coagulopathy of hemorrhagic shock is a major component of the 'lethal triad' seen in hemorrhaging patients (in conjunction with acidosis and hypothermia). The lethal triad has a very high mortality rate (over 70%) with limited ability of physicians to treat it. Evidence supporting this argument has primarily come from the conflicts in Central Asia. Several retrospective studies have been published by the US Army Institute of Surgical Research that have not only challenged this practice but have resulted in changes in how the US armed forces manage trauma patients. The US military now uses plasma in a 1:1 ratio in their traumatized soldiers (i.e. 1 unit of plasma given for every unit of packed RBC).

Major hemorrhagic injuries in non-military situations consist primarily of traumatic injuries and major blood vessel (i.e. vascular) injuries. Although all of these injuries or problems are not exactly the same as military casualties, there are major commonalities between these population groups that allow the results of the military studies to be applicable to these civilian populations. Retrospective and case-control trials in non-military trauma and in ruptured abdominal aortic aneurysms (AAA) offer indirect evidence to support a different plasma transfusion practice that is more akin to the military recommendations. Computer simulations to model massive blood transfusion scenarios also gives credence to the premise that traditional transfusion practice is incorrect for actively hemorrhaging patients and advocates the earlier use of plasma.

A retrospective chart review of 5 years of the perioperative management of Priority 1 AAA ruptures at The Ottawa Hospital was conducted with research ethics board approval. Of 145 reviewed cases, there was a 64% survival rate. The use of plasma occurred in over 75% of patients and over 99% of patients were exposed to allogeneic blood products. Plasma use was associated with poor outcomes and served as a marker for cases with higher blood loss and blood product exposure. The use of plasma was however consistent with the present recommendations and thus appeared to be reactive in nature, rather than proactive use.

A definitive trial that assesses the role of early plasma has not been performed. Unfortunately, a study to determine the full impact of an altered plasma transfusion practice would require thousands of patients. The emergency nature of these surgical patients would also make the ability to randomize patients challenging. The goal of the present trial will therefore be to assess the feasibility of such a trial. We need to assess the ability to randomize patients, to prepare plasma and deliver it in a timely fashion. Further, the logistics of having physicians to administer the study fluid (i.e. plasma or colloid control) in a timely fashion will be determined. Finally, the ability to accurately measure outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Priority 1 life-saving surgery for hemorrhagic shock due to ruptured AAA or trauma
2. Over 18 years of age

Exclusion Criteria:

1. They will not receive any blood products for religious reasons
2. If surgery is not for hemorrhagic shock (e.g. subdural evacuation)
3. Plasma already administered for documented coagulation deficit (e.g. coumadin, hemophilia)
4. Allergy to plasma (e.g. IgA deficiency) or known allergy to Voluven® solution
5. Shock that is solely due to non-hemorrhagic reasons
6. Allergy to any vitamin
7. Vital signs absent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible participants who were recruited and randomized to full participation in trial as a measure of future success completion of a larger multicenter trial. | 24 hours
  The ability to randomize patients and have them receive AB+ plasma or colloid control early in their emergency surgery.

SECONDARY OUTCOMES:
Allogeneic blood product exposure rate | Up to 24 weeks (initial hospitalization period)
  The total allogeneic blood product exposure will be recorded.
Coagulation Status and Measures | First 48 hours (initial postoperative period)
  The postoperative coagulation tests and presence/absence of a coagulopathy as measured by laboratory investigations and clinical correlation will be recorded and assessed.
Blood Loss | First 24 hours
  The total intraoperative blood loss will be recorded and any measurable blood loss from drains in the first 24 hours will also be recorded.
Transfusion Complications | Up to 24 weeks (initial hospitalization period)
  We will measure outcomes that are or potentially related to blood product transfusions including TRALI, infections, transfusion reactions, thrombotic complications, organ failure(s) and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: David T Neilipovitz, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada